CLINICAL TRIAL: NCT07147504
Title: A Retrospective Study on the Relationship Between Mortality Rates of Fractures in Different Sites and Factors Such as Age, Metabolism, and Nutritional Status in Elderly Patients: A Single-center Retrospective Study
Brief Title: Relationship Between Mortality Rates of Fractures in Different Sites and Several Factors in Elderly Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Chaoyin Jiang, associate chief physician, Shanghai 6th People's Hospital
Other Study IDs: 2025-KY-231(K)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Fracture Lower Leg; Fracture Dislocation of Upper Limb Joint; Spinal Fractures
Keywords: fracture; Limb fractures; Spinal fractures; Elderly people; the old; Survival rate
MeSH Terms: conditions — Spinal Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- Upper limb fractures Group
- Lower limb fracture Group
- Spinal fractures Group
- 60-64 years old Group
- 65-69 years old Group
- 70-74 years old Group
- 75-79 years old Group
- 80 years and above Group
- Normal nutritional status Group
- Malnutrition status Group
- Overnutrition status Group
- Normal metabolism Group
- Abnormal metabolism group

SUMMARY:
Background and Purpose:

As people age, bones become weaker and break more easily. Older adults (people 60 years and older) who break bones may face serious health problems and have a higher chance of dying compared to younger people. The location of the broken bone, a person's age, and overall health may affect the chances of survival.

This study will conduct a retrospective analysis of medical records from geriatric patients who underwent surgical intervention for bone fractures at Shanghai Sixth People's Hospital between 2010 and 2019. The primary objective is to identify the key prognostic factors associated with post-operative mortality in this patient cohort.

The study will retrospectively analyze the medical records of patients who meet all of the following criteria:

Aged 60 years or older at the time of fracture diagnosis. Residents of Shanghai. Diagnosed with a fracture of the extremities (upper or lower limbs) or the spine.

Underwent surgical intervention for the diagnosed fracture.

The investigators will assess the following variables as potential prognostic factors for post-operative mortality:

Fracture Characteristics: The anatomical location of the fracture (e.g., hip, spine, upper extremity, lower extremity).

Patient Demographics: The patient's age at the time of injury. Physiological Status: Indicators of the patient's nutritional and metabolic health.

Comorbidities: The presence and severity of pre-existing medical conditions.

How investigators will do this study:

This study is designed as a retrospective cohort analysis. Data will be systematically extracted from existing patient medical records. As an observational study, it involves no new interventions or modifications to patient care. The primary endpoint is all-cause mortality, which will be assessed at 1, 3, and 5 years post-operatively to determine long-term survival rates.

Investigators will group participants by:

The location of fracture (20 different bone locations); Age (60-65, 66-70, 71-75, 76-80, and over 80 years old); Nutrition and health status.

Why This Study Matters:

The results of this study will help doctors better understand which older patients are at higher risk after breaking a bone. This information could help healthcare teams provide better care and potentially save lives by identifying patients who need extra attention and treatment.

Study Details:

This study will examine records from approximately 2000 participants; All participants already received their treatment between 2010-2019; No new treatments or procedures will be performed; Participant's privacy will be completely protected; The study will take about 14 months to complete;

This research will help improve care for older adults who experience bone fractures and may guide treatment decisions for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the National Orthopedic Center of Shanghai Sixth People's Hospital between January 1, 2010, and December 31, 2019;
* Age ≥ 60 years;
* Shanghai resident registration;
* Diagnosed with limb or spinal fractures and receiving surgical treatment at Shanghai Sixth People's Hospital.

Exclusion Criteria:

* Multiple fractures;
* Conservative treatment selected;
* Incomplete medical records.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients aged 60 years and older who underwent surgical treatment for fractures
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | From enrollment to the end of data collection at 4 months
Fracture-related mortality | From enrollment to the end of data collection at 4 months

SECONDARY OUTCOMES:
Postoperative complication rate | From enrollment to the end of data collection at 4 months
Recurrent fracture rate | From enrollment to the end of data collection at 4 months

IPD SHARING:
Plan to Share IPD: No
This study uses medical data involving patients' personal information, and making it public may violate patients' privacy.

REFERENCES:
- [Result] Sine K, Lee Y, Zullo AR, Daiello LA, Zhang T, Berry SD. Incidence of Lower-Extremity Fractures in US Nursing Homes. J Am Geriatr Soc. 2019 Jun;67(6):1253-1257. doi: 10.1111/jgs.15825. Epub 2019 Feb 27. PMID 30811581
- [Result] Oertel MJ, Graves L, Al-Hihi E, Leonardo V, Hopkins C, DeSouza K, Bhattacharya RK. Osteoporosis management in older patients who experienced a fracture. Clin Interv Aging. 2016 Aug 22;11:1111-6. doi: 10.2147/CIA.S107720. eCollection 2016. PMID 27578967
- [Result] Berry SD, Daiello LA, Lee Y, Zullo AR, Wright NC, Curtis JR, Kiel DP. Secular Trends in the Incidence of Hip Fracture Among Nursing Home Residents. J Bone Miner Res. 2020 Sep;35(9):1668-1675. doi: 10.1002/jbmr.4032. Epub 2020 May 8. PMID 32302028
- [Result] Berner JE, Ortiz-Llorens M, Fries CA, Nanchahal J, Jain A; QUINTET Collaborative. Quality of Life after Open Extremity Trauma (QUINTET) study: An international, multicentric, observational, cohort study of quality of life following lower extremity open fractures. J Plast Reconstr Aesthet Surg. 2024 Dec;99:486-493. doi: 10.1016/j.bjps.2024.10.025. Epub 2024 Oct 16. PMID 39476530
- [Result] Tarride JE, Burke N, Leslie WD, Morin SN, Adachi JD, Papaioannou A, Bessette L, Brown JP, Pericleous L, Muratov S, Hopkins RB. Loss of health related quality of life following low-trauma fractures in the elderly. BMC Geriatr. 2016 Apr 19;16:84. doi: 10.1186/s12877-016-0259-5. PMID 27093957
- [Result] Larsen P, Elsoe R. Long-term effect of lower limb fractures A national register-based cohort study with a mean of 16.7 years follow-up. Injury. 2025 Apr;56(4):112239. doi: 10.1016/j.injury.2025.112239. Epub 2025 Mar 4. PMID 40056731

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT07147504/Prot_SAP_000.pdf